CLINICAL TRIAL: NCT07397611
Title: PRE-surgical NEOadjuvant Sandwich Immunotherapy With HIF inhibiTion in Renal Cell Carcinoma (PRENEOSHIFT-RCC)
Brief Title: Pre-NEOSHIFT-RCC: Neoadjuvant HIF-Inhibitor Immunotherapy in RCC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Arcus Biosciences, Inc. (Industry)
Responsible Party: Principal Investigator, Wenxin Xu, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-595
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Renal Cell Carcinoma; Kidney Cancer; Kidney Neoplasm; Renal Carcinoma
Keywords: Renal Cell Carcinoma; Kidney Cancer; Kidney Neoplasm; Renal Carcinoma; ccRCC
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — zimberelimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A: Casdatifan (Experimental): 16 participants will be enrolled and will complete the following:
  * Baseline visit
  * Cycle 1 through 3 (21 day cycles):
    --Days 1 - 21: Predetermined dose of Casdatifan 1x daily
  * standard of care nephrectomy
  * Follow up for up to 3 years
  Interventions: Drug: Casdatifan
- Group B: Casdatifan + Zimberelimab (Experimental): * 16 participants will be enrolled and will complete the following:
  * Baseline visit
  * Cycle 1 through 3 (21 day cycles):
    * Days 1 - 21: Predetermined dose of Casdatifan 1x daily
    * Day 1: Predetermined dose of Zimberelimab
  * Standard of care nephrectomy
  * Follow up for up to 3 years
  Interventions: Drug: Casdatifan; Drug: Zimberelimab

INTERVENTIONS:
Drug: Casdatifan — HIF-2α inhibitor, tablet taken orally per protocol.
  Other Names: C21H17F4NO3S; AB521
Drug: Zimberelimab — monoclonal antibody, multi-dose vial, via intravenous (through the vein) infusion, per protocol.
  Other Names: AB122
  Arms: Group B: Casdatifan + Zimberelimab

SUMMARY:
The purpose of this study is to see whether the drug casdatifan is safe and effective either by itself or in combination with the drug zimberelimab in participants with resectable clear cell renal cell carcinoma (ccRCC).

The names of the study drugs involved in this study are:

* Casdatifan (a type of HIF-2α inhibitor)
* Zimberelimab (a type of monoclonal antibody)

DETAILED DESCRIPTION:
This is a two-arm, open-label, multicenter, randomized trial to evaluate whether the drug casdatifan is safe and effective either by itself or in combination with the drug zimberelimab in participants with resectable clear cell renal cell carcinoma (ccRCC).

Participants will be randomized into 1 of 2 study groups: Group A Casdatifan vs. Group B Casdatifan plus Zimberelimab. Randomization means a participant is placed into a study group by chance.

The U.S. Food and Drug Administration (FDA) has not approved casdatifan or zimberelimab as a treatment for ccRCC.

The research study procedures include screening for eligibility, in-clinic visits, blood tests, urine tests, Computerized Tomography (CT) scans, Magnetic Resonance Imaging (MRI) scans, or Positron Emission (PET) scans, and X-rays.

It is expected that about 32 people will take part in this research study.

Arcus Biosciences, Inc. is supporting this research study by providing the study drugs casdatifan and zimberelimab.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients age ≥ 18 years.
* Histologically confirmed diagnosis of ccRCC by a core-needle biopsy. Patients who have not had prior biopsy may undergo screening if they have suspected RCC but can only proceed to registration if ccRCC (any component) is confirmed on the pre-treatment study biopsy.
* Stage cT2 RCC with grade 4 or sarcomatoid features, ≥cT3 Nx RCC, or cTany N+ RCC disease for which partial or radical nephrectomy is planned. For clinical staging, a kidney MRI is highly preferred over a CT Abdomen.
* Participants must have measurable disease i.e. a primary renal tumor that can be accurately measured in at least one dimension as ≥10 mm (≥1 cm) with CT scan or MRI. See Section 11 (Measurement of Effect) for the evaluation of measurable disease.
* Participants must be planned for surgical resection of their primary renal tumor.
* ECOG performance status of 0-1.
* Participants must have adequate organ and marrow function, based upon meeting all of the following laboratory criteria within 14 days before first dose of study treatment:

  1. Absolute neutrophil count ≥ 1.0 × 10^9/L without granulocyte colony-stimulating factor support within 2 weeks of screening laboratory sample collection.
  2. Platelet count ≥ 100 × 10^9/L without transfusion within 2 weeks of screening laboratory sample collection.
  3. Hemoglobin ≥ 10.0 g/dL (or 6.2 mmol/L).
  4. Aspartate transaminase (AST) ≤ 2.5 × upper limit of normal (ULN)
  5. Alanine aminotransferase (ALT) ≤ 2.5 × ULN.
  6. Bilirubin ≤ 1.5 × ULN (except participants with Gilbert syndrome who must have total bilirubin < 3.0 mg/dL).
  7. Activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN.
  8. Ambulatory oxygen saturation >92% on room air at time of screening.
  9. Serum albumin ≥ 2.8 g/dl.
  10. INR ≤ 1.5.
  11. Calculated creatinine clearance ≥ 40 mL/min (≥ 0.67 mL/sec) using the Cockcroft-Gault equation:

      ---Males: (140 - age) x weight (kg)/(serum creatinine [mg/dL] × 72)

      ---Females: [(140 - age) x weight (kg)/(serum creatinine [mg/dL] × 72)] × 0.85
* No exercise-induced desaturation on a 6-minute walk test, defined as a blood oxygen saturation by pulse oximetry ≤ 88%.
* No active clinical pneumonitis at screening.
* No medical history of severe chronic obstructive pulmonary disease (COPD)
* Screening echocardiogram or MUGA scan must demonstrate a left ventricular ejection fraction (LVEF) greater than the institutional lower limit of normal (LLN).
* Negative serum pregnancy test at screening for women of childbearing potential. Female subjects are considered to be of childbearing potential unless one of the following criteria is met: permanent sterilization (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or documented postmenopausal status (defined as 12 months of amenorrhea in a woman > 45 years-of-age in the absence of other biological or physiological causes. In addition, females < 55 years-of-age must have a serum follicle stimulating hormone [FSH] level > 40 mIU/mL to confirm menopause). Note: Documentation may include review of medical records, medical examination, or medical history interview by study site staff.
* Sexually active fertile subjects and their partners must agree to use highly effective methods of contraception during the course of the study and for the following durations after the last dose of treatment (whichever is later). An additional contraceptive method, such as a barrier method (eg, condom), is required. In addition, men must agree not to donate sperm and women must agree not to donate eggs (ova, oocyte) for the purpose of reproduction during these same periods. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Through 7 days after the last dose of casdatifan and 120 days after the last dose of zimberelimab for women of childbearing potential and for men
* Ability to understand and the willingness to sign a written informed consent document.
* Ability to swallow tablets.

Exclusion Criteria:

* Any prior systemic therapy for treatment of renal cell carcinoma.
* Any radiation therapy within 4 weeks before the first dose of study treatment.
* Any clear evidence of distant metastases. Enlarged lymph nodes that are planned to be removed during nephrectomy are permitted.
* Clinical pneumonitis or concern for inflammatory lung disease at time of screening.
* Any complementary medications (eg, herbal supplements or traditional Chinese medicines) with the intention to treat the disease under study within 2 weeks before first dose of study treatment.
* Other prior malignancy active within the previous year except for locally curable cancers (>90%) that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix, breast, or Gleason 6 prostate cancer. Also, indolent malignancies, including but not limited to early-stage chronic lymphocytic leukemia and follicular lymphoma, that don't require anti-cancer treatment, could be allowed after discussion with the medical monitor.
* QTc ≥ 480 msec using Fridericia's correction (QTcF) (based on an average of triplicate recordings).
* Malabsorption condition that would alter the absorption of orally administered medications.
* Patient has had any major cardiovascular event within 6 months prior to study drug administration including but not limited to myocardial infarction, unstable angina, cerebrovascular accident, transient ischemic event, pulmonary embolism, clinically significant ventricular arrhythmias (eg, sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes) or New York Heart Association Class III or IV heart failure.
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  a. Cardiovascular disorders: i. Congestive heart failure New York Heart Association Class 2 or greater, unstable angina pectoris, serious cardiac arrhythmias (eg, ventricular flutter, ventricular fibrillation, Torsades de pointes).

ii. Uncontrolled hypertension defined as sustained blood pressure (BP) > 150 mm Hg systolic or > 95 mm Hg diastolic despite optimal antihypertensive treatment.

iii. Any history of stroke (including transient ischemic attack [TIA]), myocardial infarction, or other clinically significant ischemic event within 12 months before first dose of study treatment.

iv. Clinically significant pulmonary embolism (PE) or deep vein thrombosis (DVT) or prior clinically significant venous or non-CVA/TIA arterial thromboembolic events within 3 months before to first dose of study treatment. Thrombus felt due to tumor and not a bland thrombus is permitted.

Note: Subjects with a diagnosis of DVT/PE due to bland thrombus need to be asymptomatic and have at least 4 weeks of anticoagulation before first dose of study treatment.

v. Any history of myocarditis.

b. Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation: i. Tumors invading the GI-tract from external viscera. ii. Active and symptomatic peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, or acute pancreatitis.

iii. Acute obstruction of the bowel, gastric outlet, or pancreatic or biliary duct within 6 months unless the cause of obstruction is definitively managed and subject is asymptomatic.

iv. Abdominal fistula, gastrointestinal perforation, bowel obstruction, or intra-abdominal abscess within 6 months before the first dose. Note: Complete healing of an intra-abdominal abscess must be confirmed before the first dose of study treatment.

v. Known gastric or esophageal varices. vi. Ascites requiring drainage within 28 days prior to initiation of protocol therapy c. Autoimmune disease that has been symptomatic or required treatment with 1mg/kg of corticosteroids within the past two years from the date of randomization. Diabetes mellitus and thyroid auto-immune diseases are excluded.

d. Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of randomization. Note: Inhaled, intranasal, intra-articular, or topical steroids are permitted. Adrenal replacement steroid doses > 10 mg daily prednisone equivalent are permitted. Transient short-term use of systemic corticosteroids for allergic conditions (eg, contrast allergy) is also allowed. Corticosteroids given as short course premedication is acceptable.

* Other clinically significant disorders that would preclude safe study participation.

  1. Active infection requiring systemic treatment. Note: Prophylactic antibiotic treatment is allowed.
  2. Infection with acute or chronic hepatitis B or C with detectable viral load, human immunodeficiency virus (HIV) infection with detectable viral load or acquired immunodeficiency syndrome (AIDS)-related illness.
  3. Serious non-healing wound/ulcer/bone fracture. Note: non-healing wounds or ulcers are permitted if due to tumor-associated skin lesions.
  4. Pharmacologically uncompensated, symptomatic hypothyroidism.
  5. Moderate to severe hepatic impairment (Child-Pugh B or C).
  6. History of solid organ or allogeneic stem cell transplant.
* Major surgery (as defined in Appendix B) within 4 weeks prior to first dose of study treatment. Minor surgery (eg, simple excision, tooth extraction) within 7 days before the first dose of study treatment. Complete wound healing from major or minor surgery must have occurred at least prior to the first dose of study treatment.
* Patients who are receiving treatment with strong CYP3A4 inhibitors and inducers should have a washout period of 28 days or 5 half-lives of the concerning medicine prior to starting casdatifan.
* History of psychiatric illness, mental condition or substance use disorders that are likely to interfere with ability to comply with protocol requirements or give informed consent.
* Use of any live vaccines against infectious diseases within 28 days of first dose of study drug.
* Current breastfeeding.
* Previously identified allergy or hypersensitivity to components of the study treatment formulations.
* Any use of supplemental or intermittent oxygen therapy.
* Other conditions, which in the opinion of the Investigator, would compromise the safety of the patient or the patient's ability to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Tumor Size Reduction Rate | Disease assessment will occur at pre-surgery visit week 11 ± 2 weeks.
  Tumor size reduction rate is defined as the proportion of participants who achieve any decrease in the maximal dimension of the primary tumor.

SECONDARY OUTCOMES:
Global Adverse Events (AE) Rate | Assessed from treatment start and continuing through the first long-term follow-up visit at 3 months post-surgery, for a total maximum duration of approximately 24 weeks.
  The global AE rate is defined as the proportion of participants experiencing at least one adverse event of Grade ≥2 (as Grade 1 AEs are not collected per protocol) during the protocol-specified AE reporting period. All AEs are included regardless of treatment attribution. All AEs will be defined and graded according to the National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0.
Treatment Related Adverse Events (TRAEs) Rate | Assessed from treatment start and continuing through the first long-term follow-up visit at 3 months post-surgery, for a total maximum duration of approximately 24 weeks.
  The TRAEs rate is the proportion of participants experiencing Grade ≥2 AEs that are at least possibly related to the study treatment (i.e., possibly, probably, or definitely related) during the protocol-specified AE reporting period. All AEs will be defined and graded according to the National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Wenxin Xu, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu